CLINICAL TRIAL: NCT01832922
Title: A Dose-Ranging Study of Bendamustine and Rituximab in Chronic Lymphocytic Leukemia (CLL) Patients With Comorbidities and/or Renal Dysfunction
Brief Title: BR in Patients With CLL With Comorbidities and/or Renal Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lionel.D.Lewis, MD, Professor of Medicine and of Pharmacology and Toxicology, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D13067; 3P30CA023108-31S4 (NIH)
Record Dates: First submitted 2013-04-12; First posted 2013-04-16 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: bendamustine; rituximab; Chronic Lymphocytic Leukemia; comorbidities; renal insufficiency
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Renal Insufficiency | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Significant Comorbidiities (Experimental): Significant comorbidities as defined by Cumulative Illness Rating Score (CIRS) of ≥7.
  Interventions: Drug: Bendamustine; Drug: Rituximab
- Significant renal dysfunction (Active Comparator): Significant renal dysfunction defined as CrCL 15-40 mL/min, but not receiving dialysis.
  Interventions: Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine
  Other Names: Treanda
Drug: Rituximab
  Other Names: Rituxan

SUMMARY:
This is a non-randomized, open label, dose-ranging study of Bendamustine and Rituximab (BR) in patients with previously untreated or relapsed/refractory Chronic Lymphocytic Leukemia (CLL) who have multiple comorbidities with or without renal insufficiency. These agents are FDA approved for this indication. However, full dose bendamustine is associated with significant hematologic toxicity and a high rate of infectious complications in "unfit" patients and patients with significantly impaired renal function. This study will attempt to optimize and define adequate and safe treatment protocols for these patients with comorbidities and/or renal dysfunction.

The study will accrue two independent patient cohorts which will follow a standard Phase I design. Patients with CLL who have significant comorbidities with or without minor renal dysfunction (CrCL>40 mL/min) will be accrued onto Cohort 1 of the study. Patients with significant renal dysfunction (CrCL<40 mL/min) will be accrued onto Cohort 2. Once the maximum tolerated dose (MTD) is determined, two expansion cohorts will be enrolled.

There will be a treatment period of up to six 28-day cycles. On C1D1 all qualifying patients will provide samples for biomarker analysis. Six patients without renal dysfunction and 6 to 9 patients with renal dysfunction will also provide samples for bendamustine PK analysis.

Accrual of both patient cohorts will occur simultaneously and will take place at two centers: Norris Cotton Cancer Center (NCCC) and Dana-Farber Cancer Institute (DFCI). Coordination of accrual to the study cohorts will be centralized at NCCC by Dr. Alexey V. Danilov.

DETAILED DESCRIPTION:
This is a non-randomized open label dose-ranging study of Bendamustine and Rituximab (BR) in patients with previously untreated or relapsed/refractory CLL who have multiple comorbidities (Cumulative Illness Rating Scale [CIRS]≥7) with or without renal insufficiency (estimated creatinine clearance [CrCL] 15-40 mL/min, but not receiving dialysis).

The study will accrue two independent patient cohorts. Both cohorts will follow a standard 3+3 Phase I design. Once the maximum tolerated dose (MTD) is determined, two expansion cohorts will be enrolled. Dose limiting toxicities (DLT) will be assessed during the 1st cycle of treatment.

Patients with CLL who have significant comorbidities (CIRS≥7; at least one category grade 3-4), with or without minor renal dysfunction (CrCL>40 mL/min) will be accrued onto Cohort 1 of the study. At dose level 1, patients will receive bendamustine 45 mg/m2 in combination with rituximab (375 mg/m2 with cycle 1 and 500 mg/m2 with subsequent cycles). If safe, the dose of bendamustine will be escalated to 70 mg/m2 (dose level 2). By contrast, dose de-escalation to 25 mg/m2 (dose level -1) will occur in this cohort if DLT's are encountered at dose level 1. Once an MTD is determined an expansion cohort will be accrued at that dose level to allow assessment of DLT's during subsequent cycles.

Because bendamustine has not been formally studied in patients with renal failure and due to the potential for increased frequency of toxic events in such patients, patients with significant renal dysfunction (CrCL 15-40 mL/min, but not receiving dialysis) will be accrued on Cohort 2. DLT's in 0/3 (or ≤1/6) subjects with renal dysfunction at dose level 1 (as above) will permit continued accrual of such subjects onto the expansion cohort (N=10). If unacceptable toxicity is encountered, bendamustine dose will be reduced to 25 mg/m2 (dose level -1), followed by an expansion cohort if safe (10 patients). Dose escalation will not be allowed in this cohort.

Accrual of both patient cohorts will occur simultaneously (see Schema) and will take place at two centers: the ambulatory Hematology Clinics at the Norris Cotton Cancer Center (NCCC) at Dartmouth-Hitchcock Medical Center (DHMC), Lebanon, NH (Lead [Dartmouth] Principal Investigator [Lead PI] - Alexey Danilov M.D., Ph.D.), and the CLL Center at Dana-Farber Cancer Institute (DFCI), Boston, MA (DFCI Principal Investigator [DFCI PI] - Jennifer Brown M.D., Ph.D.). Coordination of accrual to the study cohorts will be centralized at the Norris Cotton Cancer Center/DHMC by Dr. Alexey V. Danilov.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or flow cytometry confirmed diagnosis of B-cell chronic lymphocytic leukemia/small lymphocytic lymphoma (B-CLL/SLL) according to NCI-WG 1996 guidelines (41). The malignant B cells must co-express CD5 with CD19 or CD20. Patients who lack CD23 expression on their leukemia cells should be examined for (and found NOT to have) either t(11;14) or cyclin D1 overexpression, to rule out mantle cell lymphoma.
2. Active disease meeting at least 1 of the following IWCLL 2008 criteria for requiring treatment:

   1. A minimum of any one of the following constitutional symptoms:

      1. Unintentional weight loss >10% within the previous 6 months prior to screening.
      2. Extreme fatigue (unable to work or perform usual activities).
      3. Fevers of greater than 100.5 F for ≥2 weeks without evidence of infection.
      4. Night sweats without evidence of infection.
   2. Evidence of progressive marrow failure as manifested by the development of, or worsening of anemia or thrombocytopenia.
   3. Massive (ie, >6 cm below the left costal margin), progressive or symptomatic splenomegaly.
   4. Massive nodes or clusters (ie, > 10 cm in longest diameter) or progressive lymphadenopathy.
   5. Progressive lymphocytosis with an increase of >50% over a 2-month period, or an anticipated doubling time of less than 6 months.
   6. Autoimmune anemia or thrombocytopenia that is poorly responsive to corticosteroids.
3. Prior treatment: Patients have not had prior treatment of CLL OR Previously treated relapsed CLL patients must have received not more than 3 prior therapies for CLL. Prior bendamustine and rituximab are allowed.
4. Patients must have ECOG performance status 0-3.
5. Patients must have a Cumulative Illness Risk Score [CIRS]≥7 with at least one grade 3-4 category [CLL will not be considered a comorbidity]; or estimated creatinine clearance (CrCL) using the Cockcroft-Gault equation ≥15 mL/min but ≤40 ml/min (Appendix 1: CCI Criteria).
6. Patients must have organ function as defined below:

   * direct bilirubin ≤2 X institutional ULN (unless due to known Gilbert's syndrome or compensated hemolysis directly attributable to CLL)
   * AST or ALT < 2.5 X institutional ULN
   * estimated CrCL using the Cockcroft-Gault equation ≥15 mL/min.
   * Absolute neutrophil count (ANC) ≥500/mm3 independent of growth factor support;
   * platelets ≥30,000/mm3 independent of transfusion support with no active bleeding.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Women of childbearing potential must have a negative serum human chorionic gonadotropin or urine pregnancy test at screening.
9. All patients of reproductive potential (heterosexually active men and women) must agree to a use of a barrier method of contraception and a second method of contraception and men must agree not to donate sperm during the study and for 3 months after receiving the last dose of study treatment.

Exclusion Criteria:

1. Recent therapeutic intervention including a) prior nitrosoureas or mitomycin C within 6 weeks; b) therapeutic anticancer antibodies (including rituximab) within 4 weeks; c) radio- or toxin-immunoconjugates within 10 weeks; d) all other chemotherapy, radiation therapy within 3 weeks prior to initiation of therapy.
2. Inadequate recovery from adverse events related to prior therapy to grade ≤1 (excluding Grade 2 alopecia and neuropathy).
3. Bendamustine-refractory (no response to a regimen containing bendamustine) or relapse following treatment with a bendamustine-containing regimen within 6 months of treatment with that regimen.
4. Chronic use of corticosteroids in excess of prednisone 20 mg/day or its equivalent or chronic use of other immunosuppressive agents (azathioprine, methotrexate, tacrolimus, cyclosporine). Stem cell transplant recipients must have no evidence of active graft-versus-host disease.
5. History of prior malignancy except: a) Malignancy treated with curative intent and no known active disease present for ≥ 2 years prior to initiation of therapy on current study; b) adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; c) adequately treated in situ carcinomas (eg, cervical, esophageal, etc.) without evidence of disease; d) asymptomatic prostate cancer managed with "watch and wait" strategy.
6. Uncontrolled immune hemolysis or thrombocytopenia (positive direct antiglobulin test in absence of hemolysis is not an exclusion).
7. Known Richter's transformation.
8. Advanced renal failure (estimated CrCL < 15 mL/min) or on dialysis.
9. Human Immunodeficiency Virus (HIV) or Hepatitis C antibody positivity, or active hepatitis B.
10. Major surgery (requiring general anesthesia) within 30 days prior to initiation of therapy.
11. Uncontrolled bacterial, viral, or fungal infection.
12. Inability to adhere to the study schedule or the required follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04-27 (Actual); Study Completion 2016-11-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | within the first 30 days of treatment
  To evaluate the safety (MTD) of bendamustine in combination with rituximab in patients with CLL who have multiple comorbidities and/or significant renal dysfunction.

SECONDARY OUTCOMES:
tumor response to treatment | 3 years
  To evaluate the efficacy of BR in patients with CLL who have multiple comorbidities and/or significant renal dysfunction.

OTHER OUTCOMES:
plasma bendamustine concentration versus time | Days 1 and 2
  To determine the pharmacokinetic (PK) disposition of reduced dose bendamustine in patients with renal dysfunction (CrCL≤40 mL/min).
biomarker levels at baseline | prior to Day 1
  To assess whether established biomarkers (chromosomal abnormalities, immunoglobulin heavy chain [IGHV] mutational status, ZAP-70 and CD38 expression; p53 mutational status, microRNA expression profile) predict response to BR chemoimmunotherapy in patients with CLL who have significant comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire